CLINICAL TRIAL: NCT04341194
Title: Parents as Pain Management in Swedish Family-centred Neonatal Care. A Mixed Methods Approach
Brief Title: Parents as Pain Management in Swedish Neonatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Värmland County Council, Sweden (Other Government)
Collaborators: Region Örebro County (Other); Uppsala County Council, Sweden (Other Government); Dalarna County Council, Sweden (Other); Sykehuset Telemark (Other Government); Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Alexandra Ullsten, Principal Investigator, Värmland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LIVFOU-930025
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Infant Pain Management; Parent-driven Pain Management
Keywords: Infants; parents; neonatal intensive care; pain management; skin-to-skin contact; breastfeeding; live parental lullaby singing; PKU screening; participatory action research; randomized controlled trial
MeSH Terms: conditions — Agnosia; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Opaque sealed envelopes. which are randomly picked out before the meeting with each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care with glucose (No Intervention): Control Group with standard care comprises facilitated tucking done by a nurse or the parent, oral glucose (300 mg/ml) and the opportunity to suck on a pacifier or on a parent's or a nurse's plastic gloved finger. The infant is placed on an examination table for the venipuncture.
- Skin-to-skin contact (Experimental): Skin-to-skin contact is a method widely used in neonatal care globally. The infant is placed naked (except for a diaper and possibly a hat) on the parents' bare chest.
  Interventions: Behavioral: Parent-driven pain management with skin-to-skin contact
- Skin-to-skin contact/breastfeeding/parental singing (Experimental): Parent-driven interventions are skin-to-skin care, breastfeeding and multi-sensory stimulation like vocalisation. They are all a combination of multiple sensory inputs comprising auditory, tactile and olfactory recognition. Research has started to investigate breastfeeding in combination with Kangaroo-mother- care for example, which has shown to be an effective mix. A multimodal approach that includes a combination of non-pharmacological approaches is considered more effective during venipuncture than single strategies and provides greater pain relief.
  Interventions: Behavioral: Parent-driven pain management with skin-to-skin contact/breastfeeding/parental singing

INTERVENTIONS:
Behavioral: Parent-driven pain management with skin-to-skin contact — The infant is placed naked (except for a diaper and possibly a hat) on the parents' bare chest.
  Arms: Skin-to-skin contact
Behavioral: Parent-driven pain management with skin-to-skin contact/breastfeeding/parental singing — Live parental infant-directed lullaby singing is an individually tailored, non-verbal, multisensory, multimodal and affective tool to regulate the infant before, during and after venipuncture. Direct breast-feeding has demonstrated efficacy that is equal to, or greater than, sweet taste interventions in reducing behavioral and physiological responses to pain in full-term infants undergoing venipuncture with no demonstrated adverse outcomes. Direct breast-feeding should be considered the preferred first-line analgesic intervention for painful procedures performed on full-term infants.
  Arms: Skin-to-skin contact/breastfeeding/parental singing

SUMMARY:
Parents are a valuable but underused resource in neonatal pain management. In the Nordic countries, family-centred neonatal care has come a long way in welcoming and including parents in the everyday care of their infant. Nonseparation of parents and infants is a protective measure in decreasing stress in both parents and infants and should also be applicable during painful procedures. Sick newborn infants and infants that are born premature are cared for in neonatal intensive care units (NICUs). Because of the intense nature of the care the infants are subjected to an extensive amount of painful procedures and treatments needed for survival. Research shows that infants cared for in the NICU, experience on average between 7 and 17 painful procedures per day, and far from all infants receive adequate pharmacological or non-pharmacological analgesia during the procedures. The parents' role in the pain experience of older children has received considerable attention in research, but parents' participation in infant pain management has quite recently become a focus for research in nursing pain science with currently a handful studies. Research shows for example that when parents are present, the documentation of nursing pain assessment increases as well as the use of non-pharmacological pain-relieving methods, and parental presence can reduce the child's pain intensity and behavioural distress. There is no previous research within Swedish health care context that has investigated the parents' attitudes towards being involved in their infant's pain management, nor any research that previously has assessed the efficacy of combined parent-driven pain management such as skin-to-skin contact or breastfeeding including parental live lullaby singing. The objectives for the study are to investigate parents' and health professional's attitudes, experiences and perspectives on non-pharmacological parent-driven pain management and also to test the efficacy of combined parent-driven pain management such as skin-to-skin contact, breastfeeding and parental live lullaby singing.

DETAILED DESCRIPTION:
Study design and eligibility criteria:

The study design for the qualitative part of this study, tier one, is inspired by Participatory Action Research (PAR), involving both parents and health professionals in neonatal intensive care in a collaborative research project. Our ambition with the PAR design is to democratize the research process and include also the parents in the knowledge making. One focus group per region is recruited by the researchers and the participants are recruited based on their interest for parent-driven pain management. The focus groups contain two parents of infants who currently are admitted to the NICU, one parent who previously experienced NICU care, two health professionals and two researchers. In the focus groups, the NICU parents, the health professionals and the researchers will sit together discussing and sharing knowledge about parent-driven pain management interventions. The parents in the groups will then test the parent-driven interventions during a routine blood sample.The feedback from the focus groups will purportedly bring about guidelines for parent-driven pain management which are context sensitive and tailored to the Swedish family-centered NICU situation and public health care system as well as bring forth information how to implement parent-driven methods.

The second tier of the study is a randomized controlled trial. A written informed consent is acquired from each and one of the infant's parents. Healthy, full term infants who will be screened with the routine phenylketonuria (PKU) test and their parent, are enrolled and randomized into one of three groups; one control group with glucose (n= 75), one group with skin-to-skin contact (n= 75), and one group where the skin-to-skin contact is combined with breastfeeding and live parental lullaby singing (n= 75). All infants will receive effective pain management of some kind. Infants treated with sedatives or analgesics within the last 24 hours are excluded.

ELIGIBILITY:
Inclusion Criteria:

Healthy, full term infants who will be screened with the routine PKU test and their parent.

Exclusion Criteria:

Infants treated with sedatives or analgesics within the last 24 hours.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pain in infants | Through study completion, an average of 1 year.
  The primary outcome in the randomized controlled trial is pain in infants measured with the Premature Infant Pain Profile Revised (PIPP-R). The PIPP-R evaluates three behavioral facial actions (brow bulge, eye squeeze and nasolabial furrow), two physiological items (heart rate, transcutaneous oxygen saturation), and two contextual items (gestational age and behavioral state). The PIPP is weighted for younger gestational age and sleep state. Scores can range from 0 to 21, and a difference of two points between conditions can be considered clinically important.

SECONDARY OUTCOMES:
Changes in galvanic skin response | Through study completion, an average of 1 year.
  Changes in galvanic skin response (GSR), which is obtained via three electrodes on the infant's foot.
Parental rating of the infant's pain | Through study completion, an average of 1 year.
  Visual analogue scale (VAS). The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse populations.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Change in heart rate | Through study completion, an average of 1 year.
  For measuring heart rate variability.
Change in transcutaneous oxygen saturation | Through study completion, an average of 1 year.
  Changes in transcutaneous oxygen saturation, which is obtained via an electrode on the infant's foot.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Ullsten, PhD, Principal Investigator — Värmland County Council, Sweden
Locations (4):
- Sweden (4):
  - Neonatalavdelningen Centralsjukhuset i Karlstad, Karlstad, Värmland County
  - BB Falun Region Dalarna, Falun
  - Neonatalavdelningen, avd. 35, UniversitetssjukhusetX, Örebro
  - Intensivvårdsavdelningen för nyfödda, avd 95F, Akademiska barnsjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Misic MC, Ericson J, Eriksson M, Olsson E, Ullsten A. Effect of combined skin-to-skin contact, breastfeeding, and parents' live lullaby singing on relieving acute procedural pain in neonates (SWEpap): a multicenter randomized controlled trial in Sweden. BMC Pediatr. 2025 Dec 10;26(1):37. doi: 10.1186/s12887-025-06393-y. PMID 41366329
- [Derived] Olsson E, Carlsen Misic M, Dovland Andersen R, Ericson J, Eriksson M, Thernstrom Blomqvist Y, Ullsten A. Study protocol: parents as pain management in Swedish neonatal care - SWEpap, a multi-center randomized controlled trial. BMC Pediatr. 2020 Oct 12;20(1):474. doi: 10.1186/s12887-020-02356-7. PMID 33046026